CLINICAL TRIAL: NCT05253118
Title: Phase II Study of Tislelizumab Plus Pemetrexed in Patients With Relapsed or Refractory Primary Diffuse Large B-cell Lymphoma (DLBCL) of the Central Nervous System (CNS)
Brief Title: Relapsed or Refractory Primary Diffuse Large B-cell Lymphoma (DLBCL) of the Central Nervous System (CNS)
Acronym: SPECTRUM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Gyeongsang National University Hospital (Other); Kyunghee University Medical Center (Other); Inje University Haeundae Paik Hospital (Other); Chungnam National University Hospital (Other)
Responsible Party: Principal Investigator, Tae Min Kim, Principal investigator, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPECTRUM
Record Dates: First submitted 2022-02-06; First posted 2022-02-23 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: DLBCL
Keywords: DLBCL; Tislelizumab; Pemetrexed; relapsed or refractory primary diffuse large B-cell lymphoma; R/R primary DLBCL
MeSH Terms: conditions — Recurrence | interventions — tislelizumab; Pemetrexed

STUDY DESIGN:
Intervention Model Description: Tislelizumab (BGB-A317) 200mg will be administered on Day 1 of each 21-day cycle (once every 3 weeks) in combination with pemetrexed. And pemetrexed 500 mg/m2 will be administered on Day 1 of each 21-day cycle (once every 3 weeks).
Masking Description: open
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Tislelizumab (BGB-A317) 200mg will be administered on Day 1 of each 21-day cycle (once every 3 weeks) in combination with pemetrexed. And pemetrexed 500 mg/m2 will be administered on Day 1 of each 21-day cycle (once every 3 weeks).
  Interventions: Drug: Tislelizumab; Drug: Pemetrexed

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab (BGB-A317) 200mg will be administered on Day 1 of each 21-day cycle (once every 3 weeks) in combination with pemetrexed.
  Other Names: BGB-A317
Drug: Pemetrexed — Pemetrexed 500 mg/m2 will be administered on Day 1 of each 21-day cycle (once every 3 weeks).

SUMMARY:
Relapsed or refractory primary DLBCL of the CNS

DETAILED DESCRIPTION:
This is a multi-center, open label, single arm, phase 2 study designed to evaluate efficacy and safety of tislelizumab (BGB-A317) in combination with pemetrexed in patients with R/R primary DLBCL of the CNS. Twenty-eight patients will be enrolled. Eligible participants will receive combination treatment until disease progression, unacceptable toxicity, or withdrawal of informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent and can understand and agree to comply with the requirements of the study and the schedule of assessments
2. Age of 19 years or older on the day of signing the informed consent form (or the legal age of consent in the jurisdiction in which the study is taking place)
3. Histologically confirmed primary DLBCL of the CNS in the local lab
4. Relapsed or refractory disease with failure to at least one line of chemotherapy including high-dose methotrexate-containing regimen
5. At least one bi-dimensionally measurable lesion per IPCG response criteria Note: A lesion in an area subjected to prior locoregional therapy, including previous radiotherapy, is not considered measurable unless there has been demonstrated progression after the therapy as defined by IPCG response criteria.
6. Mandatory provision of next-generation sequencing (NGS) data or formalin-fixed paraffin-embedded (FFPE) archival tissue Note: Patients should submit 2 unstained slides and at least 5 cuts of tissue in 10-μm thickness. If there is local NGS data, at least 2 unstained slides are acceptable.
7. ECOG performance status 0-2
8. Adequate organ function as indicated by the following laboratory values, ≤ 28 days prior to randomization or first dose of study drug(s)

   a. Patients must not have required a blood transfusion or growth factor support ≤ 14 days before sample collection at screening for the following: i. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L ii. Platelets ≥ 75 x 109/L iii. Hemoglobin ≥ 90 g/L (9.0 g/dL)

   b. Serum creatinine ≤ 1.5 x ULN (upper limit of normal) or estimated glomerular filtration rate (eGFR) ≥ 45 mL/min/1.73 m2 by Chronic Kidney Disease Epidemiology Collaboration equation

   c. Serum total bilirubin ≤ 1.5 x ULN (total bilirubin must be < 3 x ULN for patients with Gilberts syndrome).

   d. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 x ULN if no demonstrable liver metastases, or ≤ 5 x ULN if transaminase elevation is attributable to liver metastases
9. Females of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study, and ≥ 120 days after the last dose of study drug(s), and have a negative urine (or serum) pregnancy test ≤ 7 days before initial treatment
10. Non-sterile males must be willing to use a highly effective method of birth control and not donate/bank sperm for the duration of the study and for ≥ 120 days after the last dose of tislelizumab (a 'sterile' male is defined as one for whom azoospermia has been previously demonstrate in a semen sample examination as definitive evidence of infertility)

Exclusion Criteria:

1. Secondary CNS lymphoma
2. Primary ocular lymphoma
3. A known history of HIV infection
4. Previous treatment with pemetrexed or immunotherapy including, but not limited to anti-PD-(L)1 antibody and anti-CTLA4 antibody
5. Radiotherapy to CNS lesions within 4 weeks prior to initiation of study treatment
6. Autologous stem cell transplantation as a part of treatment for primary DLBCL of the within 90 days prior to the start of the treatment
7. Has received any chemotherapy, targeted therapy, or any investigational therapies including investigational vaccine within 14 days or 5 half-lives (whichever is shorter) of the first study drug(s) administration
8. Known hypersensitivity or intolerance to pemetrexed or tislelizumab (BGB-A317)
9. Active autoimmune diseases or history of autoimmune diseases that may relapse

   Note: Patients with the following diseases are not excluded and may proceed to further screening:
   1. Controlled Type I diabetes
   2. Hypothyroidism (provided it is managed with hormone replacement therapy only)
   3. Controlled celiac disease
   4. Skin diseases not requiring systemic treatment (e.g., vitiligo, psoriasis, alopecia)
   5. Any other disease that is not expected to recur in the absence of external triggering factors
10. Any active malignancy ≤ 2 years before the first dose of study drug(s), except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated curatively (e.g., resected basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast)
11. Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤ 14 days before the first dose of study drug(s)

    Note: Patients who are currently or have previously been on any of the following steroid regimens are not excluded:
    1. Adrenal replacement steroid (dose ≤ 10 mg daily of prednisone or equivalent)
    2. Topical, ocular, intra-articular, intranasal, or inhaled corticosteroid with minimal systemic absorption
    3. Short course (≤ 7 days) of corticosteroid prescribed prophylactically (e.g., for contrast dye allergy) or for the treatment of a non-autoimmune condition (e.g., delayed-type hypersensitivity reaction caused by contact allergen)
12. With history of interstitial lung disease, non-infectious pneumonitis or uncontrolled diseases including pulmonary fibrosis, acute lung diseases, etc.
13. With severe chronic or active infections requiring systemic antibacterial, antifungal, or antiviral therapy, including tuberculosis infection, etc.

    1. Severe infections within 4 weeks before the first dose of study drug(s), including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
    2. Received therapeutic oral or intravenous antibiotics within 2 weeks before the first drug administration
14. Patients with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers whose HBV DNA is > 20 IU/mL Note: Inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B (HBV DNA < 20 IU/mL) can be enrolled. Patient taking antiviral agents should have received it more than 2 weeks before the treatment.
15. Patients with active hepatitis C virus (HCV) Note: Hepatitis C antibody (anti-HCV) is negative or anti-HCV positive with undetectable HCV RNA (< 15 IU/mL) can be enrolled. Patient taking antiviral agents should have received it more than 2 weeks before the treatment.
16. Any major surgical procedure requiring general anesthesia ≤ 28 days before the first dose of study drug(s)
17. Any of the following cardiovascular risk factors:

    1. Cardiac chest pain, defined as moderate pain that limits instrumental activities of daily living, ≤ 28 days before the first dose of study drug(s)
    2. Pulmonary embolism ≤ 28 days before the first dose of study drug(s)
    3. Any history of acute myocardial infarction ≤ 6 months before the first dose of study
    4. Any history of heart failure meeting New York Heart Association (NYHA) Classification III or IV (Appendix 6) ≤ 6 months before the first dose of study drug(s)
    5. Any event of ventricular arrhythmia ≥ Grade 2 in severity ≤ 6 months before the first dose of study drug(s)
    6. Any history of cerebrovascular accident ≤ 6 months before the first dose of study drug(s)
    7. Uncontrolled hypertension: systolic pressure ≥ 160 mmHg or diastolic pressure ≥ 100 mmHg despite anti-hypertension medications ≤ 28 days before the first dose of study drug(s)
    8. Any episode of syncope or seizure ≤ 28 days before the first dose of study drug(s)
18. Has received any herbal medicine used to control cancer within 14 days of the first study drug(s) administration.
19. Patients with toxicities (as a result of prior anticancer therapy) which have not recovered to baseline or stabilized, except for AEs not considered a likely safety risk (e.g., alopecia, neuropathy and specific laboratory abnormalities)
20. Was administered a live vaccine ≤ 4 weeks before the first dose of study drug(s) Note: Seasonal vaccines for influenza and SARS-CoV-2 (or COVID-19) are generally inactivated vaccines and are allowed. Intranasal vaccines are live vaccines and are not allowed.
21. Underlying medical conditions (including laboratory abnormalities) or alcohol or drug abuse or dependence that, will be unfavorable for the administration of study drug(s) or affect the explanation of drug toxicity or AEs or result in insufficient or might impair compliance with study conduct.
22. Concurrent participation in another therapeutic clinical study.
23. Pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study or within 120 days after the last dose of study drug(s)
24. History or current evidence of any condition or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-08-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Through study completion, an average of 1 year
  To evaluate objective response rate (ORR) of tislelizumab (BGB-A317) plus pemetrexed in R/R primary DLBCL of the CNS

SECONDARY OUTCOMES:
Progression-free survival | Through study completion, an average of 1 year
  To evaluate progression-free survival (PFS), duration of response (DoR) and overall survival (OS) of tislelizumab plus pemetrexed in R/R primary DLBCL of the CNS
Safety and Tolerability | Through study completion, an average of 1 year
  To evaluate the safety and tolerability of tislelizumab plus pemetrexed based on National Cancer Institute Common Terminology Criteria (NCI-CTCAE) version 5.0
Overall survival | Through study completion, an average of 2 years
  The length of time from the date of the first treatment to the date of any death or last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Tae Min Kim, PhD., M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Not yet